CLINICAL TRIAL: NCT04444856
Title: Clinical Outcomes of NovoSeven® Treatment in Severe Postpartum Haemorrhage - a Retrospective Single-centre Cohort Study at the University Hospital of Bern
Brief Title: Clinical Outcomes of NovoSeven® Treatment in Severe Postpartum Haemorrhage - a Study at the University Hospital of Bern
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7711-4729; EUPAS35429 (Registry Identifier: EU PAS Register); U1111-1248-2816 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Severe Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Factor VII; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NovoSeven: Women with severe postpartum haemorrhage treated with NovoSeven
  Interventions: Drug: Eptacog alfa (activated)
- Standard of care: Women with severe postpartum haemorrhage treated with standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Eptacog alfa (activated) — The women included in the study population have been treated with NovoSeven® (eptacog alfa (activated)) according to local routine clinical practice at the discretion of the treating physician.
  Groups: NovoSeven
Other: Standard of care — The women included in the study population have been treated according to local routine clinical practice at the discretion of the treating physician.
  Groups: Standard of care

SUMMARY:
This non-interventional study will compare the clinical outcomes in women with an event of severe postpartum haemorrhage treated with NovoSeven® to clinical outcomes in women with an event of severe postpartum haemorrhage not treated with NovoSeven®. The study will be a single centre retrospective cohort study of women with an event of severe postpartum haemorrhage, defined as 1.5 L of blood loss within 24 hours of delivery, in the period of 2005-2016.

ELIGIBILITY:
Inclusion Criteria:

* Females
* sPPH, defined as continuous bleeding of more than 1500 mL within 24 hours after delivery
* Inclusion in one of the four cohorts (historical cohort 1, historical cohort 2, study cohort and new cohort)

Exclusion Criteria:

* There are no exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with severe postpartum haemorrhage (sPPH) who were treated with NovoSeven® or other standard of care
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of invasive procedures (yes/no). (Invasive procedures are defined as: uterine or iliac artery ligation, radiological arterial embolisation, uterine compression sutures, or hysterectomy.) | 20 min-24 hours following time 0
  Count of participants (yes/no)
  Time 0 definition for all endpoints:
  Timescale for matching is time (in hours and minutes) since onset of sPPH. For exposed women: Time 0 is defined as time of first administration of NovoSeven®. It occurs x minutes after onset of sPPH. For matched controls: Time 0 is derived from the matching process. It is equal to the period from onset of sPPH to time of first administration of NovoSeven® for the patient for which they are a matched control.

SECONDARY OUTCOMES:
Occurrence of thromboembolic events (yes/no) | From time 0 until 5 days after time 0
  Count of participants (yes/no)
Amount of blood products transfused | From delivery to 24 hours after time 0
  Units
Estimated blood loss | From delivery to 24 hours after time 0
  mL
Occurrence of hysterectomy (yes/no) | 20 min-24 hours following time 0
  Count of participants (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com